CLINICAL TRIAL: NCT01098331
Title: Surgery and Brachytherapy: A Randomized Evaluation. Randomized Controlled Trial of Brachytherapy Versus Radical Prostatectomy in Good Risk Prostate Cancer: A Feasibility Study
Brief Title: Implant Radiation Therapy or Surgery in Treating Patients With Prostate Cancer
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed early due to poor recruitment
Sponsor: University of Southampton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: CDR0000668741; ISRCTN88144169 (Other: ISRCTN)
Record Dates: First submitted 2010-04-01; First posted 2010-04-02 (Estimated); Last update posted 2021-12-27 (Actual); Status verified 2021-12

CONDITIONS: Prostate Cancer
Keywords: stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Brachytherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm Rx1: Radical Prostatectomy (Other): Arm Rx1: Radical Prostatectomy
  Interventions: Procedure: Radical Prostatectomy
- Arm Rx2: Brachytherapy (Other): Arm Rx2: Brachytherapy
  Interventions: Procedure: Brachytherapy

INTERVENTIONS:
Procedure: Radical Prostatectomy
  Arms: Arm Rx1: Radical Prostatectomy
Procedure: Brachytherapy
  Arms: Arm Rx2: Brachytherapy

SUMMARY:
RATIONALE: Receiving standard information and watching a video or DVD at home that describes treatment options and treatment outcomes may help patients decide to receive treatment in a clinical trial.

PURPOSE: This randomized clinical trial is studying implant radiation therapy to see how well it works compared with surgery in treating patients with prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the proportion of patients consenting to the treatment randomization of brachytherapy vs radical prostatectomy in treating patients with good-risk prostate cancer.
* Determine the feasibility of randomization, in terms of average accrual rate per center, during the last 6 months of recruitment.

Secondary

* Determine the decisional quality post-treatment in these patients.
* Determine the compliance with allocated treatment in these patients.
* Determine the clinical failure in these patients.
* Determine the PSA relapse in these patients.
* Determine the patient-reported quality of life.
* Compare the toxicity of these regimens.

OUTLINE: This is a multicenter study.

* Part 1 (decision-aid randomization): Patients are stratified according to participating center. Patients are randomized to 1 of 2 Decision-Aid arms.

  * Arm I (standard patient information): Patients receive standard patient information according to routine clinical practice and preferred materials of each center. This information typically includes booklets about prostate cancer and its treatment, contact details for sources of further information (e.g., prostate support groups, prostate charities, and web-based information), and access to a specialist nurse as required.
  * Arm II (standard patient information + decision aid): In addition to standard information as described in Arm I, patients are given a 30-minute Decision-Aid video or DVD to take home. The Decision Aid describes the standard treatment options available to patients, provides detailed information about treatment outcomes in relation to individual patient characteristics, and seeks to help patients apply their own personal values to their treatment decision. Patients may watch the audio-visual aid as many times as they wish.

Patients who decide to choose a treatment are removed from study; patients who agree to undergo treatment randomization proceed to part 2 of the study.

* Part 2 (treatment randomization): Patients are stratified according to risk (low risk vs intermediate risk). Patients are randomized to 1 of 2 treatment arms.

  * Arm I (radical prostatectomy): Patients undergo surgery within 60 days of randomization. The surgical technique for radical prostatectomy may be retropubic, transperineal, laparoscopic or robotic. Pelvic lymph node surgery is permitted at the discretion of the treating surgeon. Unilateral or bilateral nerve-sparing techniques may be used at the discretion of the treating surgeon.
  * Arm II (brachytherapy): Patients undergo brachytherapy within 60 days of randomization. Brachytherapy seeds may be implanted using pre-loaded needles or a MICK® applicator of either iodine I 125 or palladium Pd 103.

Patient-reported quality-of-life data is collected to assess erectile function, urinary function, bowel function, and general quality of life at baseline and during follow up.

Patients are followed at 1 and 4 months, every 4 months for 2 years, every 6 months for 3 years, then annually for 5 years.

Peer Reviewed and Funded or Endorsed by Cancer Research UK

ELIGIBILITY:
DISEASE CHARACTERISTICS

Meeting 1 of the following criteria:

* Prostate cancer or suspected prostate cancer confined to the prostate (Decision-Aid Randomization) Clinical stage T1/T2, Due for prostate biopsy or prostate biopsy performed in the last 6 weeks, PSA < 15 ng/mL
* Histologically confirmed prostate cancer (Treatment Randomization): Clinical stage T1/T2, Re-biopsy after a period of active surveillance is at the discretion of the treating investigator, Must meet 1 of the following risk criteria (PSA test < 3 months prior to treatment intervention), Low risk: Gleason score ≤ 6 (no tertiary grade 4 or 5) with a PSA of < 10 ng/mL, intermediate-risk: Gleason score 3 + 4 (no tertiary grade 5) with a PSA > 10 ng/mL but ≤ 15 ng/mL, Transrectal ultrasound prostate volume ≤ 50 cc

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Life expectancy > 10 years (Decision-Aid Randomization)
* Satisfactory results from biochemical and hematological profiles that, in the opinion of the investigator, does not preclude patient from the trial
* No unacceptable risk for radical prostatectomy or prostate brachytherapy
* INR < 1.5
* No severe lower urinary tract symptoms
* No significant obstructive urinary symptoms (i.e., peak urine flow rate < 10 mL per second, and/or post micturition bladder volume > 100 mL)
* No other clinical or medical condition that, in the opinion of the investigator, precludes patient from taking part in the trial
* No other active malignancy likely to interfere with subsequent protocol treatment and follow-up

PRIOR CONCURRENT THERAPY:

* No prior pelvic radiotherapy
* No prior abdominoperineal (AP) rectal excision
* No prior standard transurethral resection of prostate
* No prior or concurrent neoadjuvant or adjuvant hormonal treatment, (e.g., LHRH agonists, or anti-androgens or estrogens)
* At least 5 days since prior aspirin or clopidogrel
* No concurrent warfarin

Ages: 18 Years to 120 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male
Enrollment: 30 (Actual)
Dates: Start 2008-06-01 (Actual); Primary Completion 2013-06-01 (Actual); Study Completion 2013-06-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients consenting to the treatment randomization | 6 months
Feasibility of randomization in terms of average accrual rate per center during the last 6 months of recruitment | 6 months

SECONDARY OUTCOMES:
Compliance with allocated treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Bottomley, Principal Investigator — Leeds Cancer Centre at St. James's University Hospital
Locations (1):
- Leeds Cancer Centre at St. James's University Hospital, Leeds, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eccles BK, Cross W, Rosario DJ, Doble A, Parker C, Logue J, Little L, Stanton L, Bottomley D. SABRE 1 (Surgery Against Brachytherapy - a Randomised Evaluation): feasibility randomised controlled trial (RCT) of brachytherapy vs radical prostatectomy in low-intermediate risk clinically localised prostate cancer. BJU Int. 2013 Aug;112(3):330-7. doi: 10.1111/bju.12127. PMID 23826842